CLINICAL TRIAL: NCT05062824
Title: Pilot Testing of Baby Feed: A Web Application for Health Professionals and Parents to Improve Infant Diets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Cristina Palacios, PhD, Associate Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-20-0498
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Weight and length are being collected by the nurse in Borinquen Health Center, they are blinded to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention will have access to Baby Feed
  Interventions: Behavioral: Baby Feed
- Standard Care (No Intervention): Participants in the standard care group will NOT have access to Baby Feed

INTERVENTIONS:
Behavioral: Baby Feed — Baby Feed web portals can (1) Quickly and easily evaluate infant diet using a validated Infant Food Frequency Questionnaire (infant FFQ) developed by our group14. [Parental FFQ portal]; (2) Provide automatic results to healthcare professionals on nutrients and foods/beverages consumed above or below the recommended levels to discuss with parents for improving the infant's diet. Also, to provide recommendations for amounts of foods/beverages that the infant should be consuming by age [Clinician Portal]; (3) Give online access to parents to these diet recommendations to implement at home, with an easy tracking component [Parent's Portal].
  Arms: Intervention

SUMMARY:
This project will pilot test "Baby Feed" online web portals among clinicians and parents to learn about their experience with the portals. Baby Feed evaluates infant diets online using a validated Infant Food Frequency Questionnaire, provides immediate results online to health care providers on nutrients and foods/beverages consumed above or below the recommended levels, provides current diet recommendations by infant's age online, and helps track progress at home. The investigators will recruit 2 clinicians from Borinquen Health Care Center in Miami and 50 of their patients (parents with infants) scheduled for a routine Well-Child Visit when infants are 4-12 months old. Participants will be equally randomized to the intervention group or the control group. If randomized to Baby Feed, parents will discuss the results with the healthcare professional and track their infants' diets at home. Parents in the Control group will only complete the infant FFQ online but will not have access to the other features of Baby Feed. After 3 months, the investigators will evaluate the infant diet and weight gain during this period.

DETAILED DESCRIPTION:
This project will pilot test "Baby Feed" online web portals among clinicians and parents to learn about their experience with the portals. Baby Feed can (1) Quickly and easily evaluate infant diets online using a validated Infant Food Frequency Questionnaire (FFQ) developed by the Principal Investigator [Parental Portal]; (2) Provide immediate results online to health care providers on nutrients and foods/beverages consumed above or below the recommended levels [Clinician Portal]; (3) Provide current diet recommendations by infant's age online to health care providers to discuss with parents, with the goal of improving their infant's diet [Clinician Portal]; (4) Give online access of the infant diet recommendations to parents for home implementation, with an online short tracking component [Parental Portal].

The investigators will recruit 2 clinicians from Borinquen Health Care Center in Miami and 50 of their patients (parents with infants) scheduled for a routine Well-Child Visit when infants are 4-12 months old. Participants will be equally randomized to the intervention group or the control group. All parents will first complete the Infant FFQ online. Those randomized to Baby Feed will discuss the results as a part of the Well-Child Visit with the healthcare professional, who will also have access to the results from the Clinician Portal. They will discuss the most relevant results and the dietary recommendations to follow at home. Parents will also be able to see the recommendations online in the Parental Portal in a friendly and graphic way to follow easily at home. Parents will be prompted to complete the online short tracking questions once per week to evaluate how well they are following the dietary recommendations during the duration of the study: 3 months. Parents in the Control group will only complete the infant FFQ online but will not have access to the other features of Baby Feed. After 3 months, the investigators will evaluate the infant diet by reviewing the results from the infant FFQ at baseline and 3 months later in both groups. The investigators will also evaluate weight gain during this period and compare between groups. For this, the investigators will ask all parents to complete online a short form with the weight and length of the baby as recorded by the nurse in each Well-Child Visit at baseline and follow-up visits.

RISKS/BENEFITS: The main risk or discomfort from this research is the disclosure of personal information. The main benefit to those randomized to the intervention group is that clinicians will be receiving automatic results and dietary recommendations in "Baby Feed" online to discuss with parents, and for parents is receiving dietary recommendations from "Baby Feed" online to improve their infant's diet.

IMPORTANCE OF THE KNOWLEDGE: Baby Feed could be an important tool to help promote adherence to diet recommendations which could translate into healthy weight gain during the first year and thus prevent long-term obesity.

ELIGIBILITY:
Inclusion Criteria:

* parent/guardian responsible for infant's care;
* parent of an infant age 4 to 12 months, who is healthy and with any weight status;
* have internet access;
* willing to participate for the full study duration of 2 weeks;

Exclusion criteria:

* parents of infants with special diets, limited mobility, preterm birth of < 37 weeks, birthweight < 10th or > 90th percentile;
* parent/guardian unable to consent to participate.

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Infant's diet | 3 months
  Results from the infant FFQ will be analyzed to calculate if percentage change of the foods and beverages consumed above or below the recommended levels changed during this study period
Diet quality using the Diet Quality Index Score (DQIS) | 3 months
  Using the results from the infant FFQ, the investigators will calculate the DQIS score, which is composed of 9 food groups: breastfeeding and milk, grains, proteins, vegetables, fruits, 100% juices, sugar-sweetened beverages, sweets, and salty snacks. A total of 5 points are assigned if the intake is within the recommended amounts, 2.5 points if the intake is slightly over or under recommended amount, and 0 points if the intake is excessive or not consumed. The points are summed, and diet quality is categorized as Excellent (score: 45-55), Good (score: 35-44), Needs Improvement (score: 25-34), and Poor (score: 0-24).

SECONDARY OUTCOMES:
Rate of weight gain | 3 months
  The investigators will calculate the weight z score and weight-for-length z score using the WHO Anthro Survey Analyzer. The rate of weight gain will be calculated as the change in weight z score between visits and categorized as: (1) Adequate weight gain (change of -0.67 to 0.67 standard deviations; (2) Rapid weight gain in (change > 0.67 standard deviations); (3) Slow weight gain (change of < -0.67 standard deviations).
Parenting Self-Efficacy | 3 months
  This will be assessed using a validated questionnaire, as mediator of behavioral change. The investigators will evaluate changes in the level of confidence that parents feel about feeding their baby between baseline and follow up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Borinquen Medical Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palacios C, Bolton J, Wang W, Gatto A, Concepcion L, Sadjadi M, Varella M, Hannan J. Development and pilot testing of the Baby-Feed web application for healthcare professionals and parents to improve infant diets. Int J Med Inform. 2023 Jun;174:105047. doi: 10.1016/j.ijmedinf.2023.105047. Epub 2023 Mar 17. PMID 36948062